CLINICAL TRIAL: NCT02212639
Title: Phase II Multicentric Study of Digoxin Per os in Classic or Endemic Kaposi' s Sarcoma
Acronym: KADIG 01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130944; 2014-001741-24 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Kaposi' s Sarcoma; Classic Kaposi' s Sarcoma; Endemic Kaposi' s Sarcoma; Lymph Angio Proliferations
Keywords: Kaposi' s sarcoma; Digoxin
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digoxin (Experimental): All patients will receive Digoxin without interruption. Doses can be modified individually to reach a serum drug concentration of 0.6 to 1.2 ng/ml for patients <75 years and between 0.5-0.8 ng/ml in patients older than 75 years
  Interventions: Drug: digoxin

INTERVENTIONS:
Drug: digoxin — All patients will receive Digoxin without interruption. Doses can be modified individually to reach a serum drug concentration of 0.6 to 1.2 ng/ml for patients <75 years and between 0.5-0.8 ng/ml in patients older than 75 years

SUMMARY:
Classic and endemic Kaposi's sarcoma (KS) are lymph angio proliferations associated with human herpes virus 8 (HHV8) which treatment is poorly codified. Chemotherapies give at best 30-60% of transient responses. While interferon responses are frequent, this drug is often poorly tolerated in elderly patients. Therefore new therapies are needed. Classic KS represents an ideal model for evaluating new drugs since patients do not receive concomitant immunosuppressive regimens nor antiviral therapies.

Hypoxia-inducible factor 1(HIF-1 alpha) is a major regulator of solid tumor growth and therefore a suitable target currently explored in many cancers. Moreover HIF-1 alpha enhances HHV-8 gene expression in KS and induces lytic replication cycle. Digoxin has anti cancer effect in vivo through HIF-alpha down regulation in several preclinical tumor models including KS. The identification of HIF-1 alpha as a key factor in HHV8 replication prompt us to explore inhibition of HIF-1 alpha by digoxin as a potential therapeutic approach for KS treatment it has and consequently may down regulate HHV-8 replication in KS. This latter approach is heightened by recent data suggesting that Digoxin has some efficacy in vitro against others human herpes virus i.e. Herpes simplex and Cytomegalovirus (8) (9)

In this study the investigators shall evaluate the benefit and safety profile of digoxin in classic and endemic KS (serum drug concentration of 0.6 to 1.2 ng/ml for patients <75 years and between 0.5-0.8 ng/ml in patients older than 75 years The participants will take study drug digoxin, for a total of 6 cycles (4 weeks/cycle).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years <à 80 years
* Classic or endemic histologically confirmed Kaposi's Sarcoma (KS)
* Progressive disease
* KS with more than 10 lesions or involving more than one limb segment or with involvement >3% body surface
* KS with at least 4 lesions ≥5mm
* Patients should have at least 2 others cutaneous tumor available for repeated pharmacodynamics evaluation
* At least 4 weeks wash out for all KS specific therapies including chemotherapy and immunotherapy
* Signed informed consent

Exclusion Criteria:

* Symptomatic visceral lesions
* Eastern Cooperative Oncology Group ( ECOG) performance status > 1
* Life expectancy of ≤ 6 months
* Patients already receiving digoxin
* hepatic dysfunction defined as serum bilirubin>25 µm/l, transaminases > 3.0 times the upper limit of normal (ULN) (5ULN in cases of liver metastases)
* bone marrow dysfunction defined as absolute neutrophil count<1500/mcl, platelets<150000/mcl or hemoglobin<8g/dL
* renal failure with creatinine clearance< 40ml/mn
* HIV positive, active infectious hepatitis, type A, B or C
* Uncontrolled systemic infection
* Pregnant or lactating women
* Presence of any of the following on electrocardiogram (ECG): atrial arrhythmias, including atrial fibrillation and flutter with Wolff-Parkinson-White syndrome; auricular ventricular (AV) block; heart rate < 60 beats/minute and > 100 beats/minute; ventricular fibrillation; ventricular tachycardia; premature ventricular contractions.
* History of or current cardiac arrythmia including sinus node disease, history of AV Block, accessory AV pathway (Wolff-Parkinson-White Syndrome), history myocardial infarction, any significant valvulopathy.
* Electrolyte imbalance (hypokalemia, hypo- or hypercalcemia, hypomagnesemia)
* Severe pulmonary disease and hypoxia
* Medical conditions such as uncontrolled hypertension, uncontrolled diabetes mellitus, hypothyroidism or hyperthyroidism, which would, in the opinion of the investigator, make this protocol unreasonably hazardous.
* Major thoracic or abdominal surgery within the prior 3 weeks.
* GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Immunosuppressive regimen should not be allowed including corticosteroids
* Use of any prohibited concomitant medications:

  * the calcium channel blockers diltiazem or verapamil;
  * Class I and III cardiac arrhythmic agents (such as quinidine, amiodarone);
  * beta-blockers (such as atenolol, metoprolol);
  * indomethacin (Indocin);
  * calcium carbonate antacids (e.g., Maalox, Tums, Rolaids);
  * Calcium
  * omeprazole;
  * antidiarrheal adsorbents (kaolin and pectin);
  * antibiotics P450 inhibitors clarithromycin, erythromycin telithromycin and other P450 inhibitors./such as Ritonavir)
* Persistent Grade >2 treatment-related toxicity from prior therapy
* History of any digoxin-related or drug induced anaphylactic reaction
* Use of any other investigational agent
* Patient without health insurance coverage
* Patient under guardianship
* Enrollment into a clinical trial within last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
tumor response | at 3 months
  The primary endpoint will be tumor response, at 3 months. Assessed by AIDS Clinical Trials Group (ACTG) criteria ;Complete response (CR) will be defined as the absence of detectable residual disease lasting for at least 4 weeks; patients whose only remaining manifestation of KS are pigmented macules could be classified as having had a complete response if malignant cells are absent on biopsy of at least one lesion. Patients with visceral disease on entry who have complete resolution of cutaneous lesions as described above could be considered to have a CR only if no residual disease was detected on endoscopic or radiographic restaging.

SECONDARY OUTCOMES:
Best overall response during the trial | at 6 months
  Best overall response during the trial, defined by the best response recorded from the start of treatment until disease progression/recurrence or treatment interruption for any reason
Response rate at 6 months | at 6 months
number of lesions | at 3 months
  number of lesions
size of target lesions | at 3 months
tumor infiltration of target lesions | at 3 months
lymphedema | at 3 months
  lymphedema (scale of 0 (absence)-3 (painful or oozing), circumference)
Time to response | at 3 months
Time to progression | at 3 months
toxicity | at 6 months
  Safety and tolerance aspects, they will be assessed in terms of drug toxicity evaluated by clinic and on laboratory parameters and scored according Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: celeste lebbe, MDPHD, Principal Investigator — APHP
Locations (1):
- Saint-Louis Hospital, Paris, France